CLINICAL TRIAL: NCT01635933
Title: A Comparison of a Colored Silicone Hydrogel Lens Versus a Colored HEMA Lens
Brief Title: A Comparison of AIR OPTIX® COLORS Versus FRESHLOOK® COLORBLENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: C-12-005
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Myopia
Keywords: contact lenses; color contact lenses; myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX® COLORS (Experimental): Lotrafilcon B contact lens with color worn in daily wear modality for 4 weeks. Lenses were worn bilaterally for a minimum of 5 days per week, 8 hours per day.
  Interventions: Device: Lotrafilcon B contact lens with color
- FRESHLOOK® COLORBLENDS (Active Comparator): Phemfilcon A contact lens with color worn in daily wear modality for 4 weeks, with a replacement pair dispensed at 14 days. Lenses were worn bilaterally for a minimum of 5 days per week, 8 hours per day.
  Interventions: Device: Phemfilcon A contact lens with color

INTERVENTIONS:
Device: Lotrafilcon B contact lens with color — Silicone hydrogel contact lens with color.
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX® COLORS
Device: Phemfilcon A contact lens with color — Hydrogel contact lens with color.
  Other Names: FRESHLOOK® COLORBLENDS
  Arms: FRESHLOOK® COLORBLENDS

SUMMARY:
The purpose of this study was to evaluate the overall comfort of AIR OPTIX® COLORS compared to FRESHLOOK® COLORBLENDS in habitual wearers of the FRESHLOOK® COLORBLENDS .

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign the Informed Consent document. If under legal age of consent, legally authorized representative must sign also Informed Consent document.
* Able to achieve visual acuity of at least 20/30 (Snellen) in each eye at distance with contact lenses and best corrected visual acuity (BCVA) ≥ 20/25 in each eye.
* Manifest cylinder less than or equal to 0.75 diopters (within the previous year) in each eye.
* Successful wear of FRESHLOOK® COLORBLENDS spherical soft contact lenses in both eyes (in the protocol-specified colors) during the past three months for a minimum of 5 days per week and 8 hours per day.
* History of at least 5 days of successful use with both lenses (minimum of 8 hours/day) of one of the protocol-specified lens care solutions/multi-purpose solutions (MPS).
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the test articles or affect the results of this study.
* Wears habitual lenses in an extended wear modality (sleeping in lenses overnight / not removing lenses on a daily basis).
* Monovision, monocular (only one eye with functional vision) or fit with only one lens.
* History of intolerance or hypersensitivity to any component of the test articles.
* Use of any over-the-counter or prescribed topical ocular medications within the previous 7 days (excluding rewetting drops).
* Moderate or severe corneal edema, corneal vascularization, corneal staining, injection, tarsal abnormalities, "other" complications; and any corneal infiltrates.
* Current or history of ocular infection, severe inflammation, or disease within previous 6 months.
* Any systemic disease (including allergies, respiratory infections or colds) that may affect the eye or be exacerbated by use of contact lenses or contact lens solutions.
* Participation in any investigational clinical study within previous 30 days.
* Other protocol-defined exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Holden Thomas, O.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 24 study centers located in the United States.
Pre-assignment Details: Of the 370 participants enrolled and randomized, 4 did not meet inclusion/exclusion criteria, 2 were lost to follow-up, and 1 declined participation. This reporting group includes all participants exposed to the study product (363).
Period: Overall Study
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Started | 178 | 185
Completed | 176 | 177
Not Completed | 2 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 5
Not completed — Subject decision | 1 | 1
Not completed — Noncompliance | 0 | 1
Not completed — No longer had transportation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population includes all participants exposed to the study product (363).
Groups:
- Total: Total of all reporting groups
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS | Total
Number analyzed (Participants) | 178 | 185 | 363
Age, Customized [Number; unit: participants]
  16-17 years | 9 | 10 | 19
  18-64 years | 167 | 174 | 341
  ≥65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 166 | 330
  Male | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Overall Comfort
Description: Overall comfort, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Day 28
Population: The analysis population includes all enrolled and dispensed participants who had at least one study visit after being dispensed with study lenses (N=178,185). No imputation was used for the missing values. Here, "n" is the number of participants with non-missing values at the specific time point for each arm group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 178 | 185
Units on a scale
  Day 14 (n=175,181) | 8.7 (1.7) | 8.6 (1.8)
  Day 28 (n=176,176) | 8.7 (1.7) | 8.5 (1.7)

2. Secondary Outcome: Subjective Rating of Overall Vision
Description: Overall vision, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 178 | 185
Units on a scale
  Day 14 (n=175,181) | 8.8 (1.6) | 8.7 (1.5)
  Day 28 (n=176,177) | 8.9 (1.5) | 8.7 (1.5)

3. Secondary Outcome: Proportion of Subjects Preferring Study Lens (Strongly or Somewhat)
Description: Participants were asked to compare the study lenses to their habitual lenses using a 5-point scale: strongly prefer study lenses, somewhat prefer study lenses, no preference, somewhat prefer habitual lenses, and strongly prefer habitual lenses, where 'study lenses' refer to either test or control depending on the treatment group. Proportion of subjects preferring study lens is reported as the percentage of participants who strongly or somewhat preferred the study lens.
Time Frame: Day 28
Population: The analysis population includes all enrolled and dispensed participants who had at least 1 study visit after being dispensed the study lenses. No imputation was used for missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 175 | 177
Percentage of participants | 54.3 | 45.2

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected for the duration of the study (3 months). AEs were obtained as solicited comments from subjects and as observations by the study Investigator as outlined in the study protocol.
Description: The analysis population includes all participants exposed to the study product. An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings), whether or not related to the investigational medical device.
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Serious Adverse Events (participants affected / at risk) | 1/178 | 2/185
Other Adverse Events (participants affected / at risk) | 0/178 | 0/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIR OPTIX® COLORS (N=178) | FRESHLOOK® COLORBLENDS (N=185)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 — Not related
Injury (Injury, poisoning and procedural complications) | 1 | 0 — Injuries due to a car accident. Not related.
Cholecystitis infective (Infections and infestations) | 0 | 1 — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.